CLINICAL TRIAL: NCT00634244
Title: A Phase II Randomized Trial of Carboplatin and Topotecan; Flavopiridol, Mitoxantrone and Cytosine Arabinoside; and Sirolimus, Mitoxantrone, Etoposide and Cytosine Arabinoside for the Treatment of Adults With Primary Refractory or Initial Relapse of Acute Myelogenous Leukemia (AML)
Brief Title: Comparing Three Different Combination Chemotherapy Regimens in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00520; NCI-2009-00520 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); E1906 (Other: ECOG-ACRIN Cancer Research Group); U10CA021115 (NIH)
Record Dates: First submitted 2008-03-11; First posted 2008-03-12 (Estimated); Results first posted 2015-07-07 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-04

CONDITIONS: Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Recurrent Adult Acute Myeloid Leukemia
Keywords: Acute Myelogenous Leukemia (AML), Carboplatin, Topotecan, Flavopiridol, Mitoxantrone, Cytosine Arabinoside, Sirolimus, Etoposide
MeSH Terms: conditions — Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute | interventions — alvocidib; Mitoxantrone; Carboplatin; Cytarabine; Sirolimus; Etoposide; Topotecan; trioctyl phosphine oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A (carboplatin and topotecan hydrochloride) (Experimental): Patients receive carboplatin and topotecan hydrochloride IV continuously over 24 hours on days 1-5.
  Interventions: Drug: carboplatin; Drug: topotecan hydrochloride
- Arm B (alvocidib, mitoxantrone, cytarabine) (Experimental): Patients receive alvocidib IV over 4.5 hours QD on days 1-3, cytarabine IV continuously over 72 hours on days 6-8, and mitoxantrone hydrochloride IV over 1-2 hours on day 9.
  Interventions: Drug: alvocidib; Drug: mitoxantrone hydrochloride; Drug: cytarabine
- Arm C (sirolimus, mitoxantrone, etoposide, cytarabine) (Experimental): Patients receive sirolimus PO QD on days 2-9, mitoxantrone hydrochloride IV over 15 minutes QD, etoposide IV over 1 hour QD, and cytarabine IV over 3 hours QD on days 4-8 or 5-9. (Closed to accrual)
  Interventions: Drug: mitoxantrone hydrochloride; Drug: cytarabine; Drug: sirolimus; Drug: etoposide

INTERVENTIONS:
Drug: alvocidib — Given IV
  Other Names: FLAVO; flavopiridol; HMR 1275; L-868275
  Arms: Arm B (alvocidib, mitoxantrone, cytarabine)
Drug: mitoxantrone hydrochloride — Given IV
  Other Names: CL 232315; DHAD; DHAQ
  Arms: Arm B (alvocidib, mitoxantrone, cytarabine); Arm C (sirolimus, mitoxantrone, etoposide, cytarabine)
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
  Arms: Arm A (carboplatin and topotecan hydrochloride)
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
  Arms: Arm B (alvocidib, mitoxantrone, cytarabine); Arm C (sirolimus, mitoxantrone, etoposide, cytarabine)
Drug: sirolimus — Given PO
  Other Names: AY 22989; Rapamune; rapamycin; SLM
  Arms: Arm C (sirolimus, mitoxantrone, etoposide, cytarabine)
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
  Arms: Arm C (sirolimus, mitoxantrone, etoposide, cytarabine)
Drug: topotecan hydrochloride — Given IV
  Other Names: hycamptamine; Hycamtin; SKF S-104864-A; TOPO
  Arms: Arm A (carboplatin and topotecan hydrochloride)

SUMMARY:
This randomized phase II trial is comparing three different combination chemotherapy regimens to see how well they work in treating patients with relapsed or refractory acute myeloid leukemia. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells. It is not yet known which combination chemotherapy regimen is more effective in treating patients with relapsed or refractory acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the complete remission (CR) + cytogenic complete remission (CRc) + morphologic complete remission with incomplete blood count recovery (CRi) rate of carboplatin and topotecan; flavopiridol, mitoxantrone and cytosine arabinoside and sirolimus, mitoxantrone, etoposide and cytosine arabinoside in adult patients with refractory or relapsed acute myeloid leukemia (AML).

NOTE: Since the CRc patients are required to be either CR or CRi, we only report the rate of CR+CRi in the results section.

II. To determine the rate of treatment failure of these regimens. III. To determine the incidence and severity of toxicities of these regimens. IV. To analyze the predictive value of blast cell properties that have been suggested to determine response. (Correlative laboratory studies) V. To determine whether pretreatment levels of B-cell chronic lymphocytic leukemia (CLL)/lymphoma 2 (Bcl-2) or, alternatively, whether a therapy-induced change in topoisomerase I levels correlates with response to this regimen. (Correlative laboratory studies) VI. To assess the impact of clonal evolution by comparing cytogenetic abnormalities at the time of relapse with those at initial diagnosis and correlating these abnormalities and changes with response to the treatment regimens in this protocol. (Cytogenetic and fluorescent in situ hybridization [FISH] studies) VII. Panel FISH studies for common AML rearrangements will be performed on relapse AML specimens to determine the presence of these recurrent AML abnormalities and to evaluate for subtle additional abnormalities consistent with clonal evolution in these relapse specimens. (Cytogenetic and FISH studies)

OUTLINE: Patients are randomized to 1 of 3 treatment arms.

INDUCTION THERAPY:

ARM A: Patients receive carboplatin and topotecan hydrochloride intravenously (IV) continuously over 24 hours on days 1-5.

ARM B: Patients receive alvocidib IV over 4.5 hours once daily (QD) on days 1-3, cytarabine IV continuously over 72 hours on days 6-8, and mitoxantrone hydrochloride IV over 1-2 hours on day 9.

ARM C: Patients receive sirolimus orally (PO) QD on days 2-9, mitoxantrone hydrochloride IV over 15 minutes QD, etoposide IV over 1 hour QD, and cytarabine IV over 3 hours QD on days 4-8 or 5-9. (Closed to accrual)

After completion of induction therapy, patients in all arms undergo bone marrow aspirate and biopsy. Patients with persistent leukemia (i.e., leukemic blasts >= 10%) are removed from study and are offered alternative therapy at the discretion of the investigator. Patients who achieve CR proceed to consolidation therapy or receive alternative therapy at the discretion of the investigator.

CONSOLIDATION THERAPY: Beginning within 2-6 weeks after documentation of CR, patients may receive up to 2 additional courses of the same treatment they received during induction therapy. Courses repeat every 4-10 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed periodically for up to 3 years.

ELIGIBILITY:
Inclusion Criteria

Induction Therapy:

* Patients must have morphologic proof (from bone marrow aspirate, smears or touch preps of marrow biopsy) of acute myelogenous leukemia (AML) with >= 10% blasts within two weeks prior to induction randomization

  * NOTE: Patients must be registered to E3903 (Ancillary Laboratory Protocol for Collecting Diagnostic Material on Patients Considered for Eastern Cooperative Oncology Group [ECOG]-American College of Radiology Imaging Network [ACRIN] Treatment Trials for Leukemia or Related Hematologic Disorders) and must undergo eligibility testing for the study by multiparameter flow cytometry
  * All immunodiagnoses are eligible for E1906, except acute promyelocytic leukemia (APL) (proven by the presence of promyelocytic leukemia (PML)/retinoic acid receptor (RAR) alpha); cases of APL can become eligible if the patient is ineligible for an ECOG-ACRIN APL trial or if all-trans retinoic acid or arsenic trioxide is not planned as part of the treatment regimen
* Patients must qualify for one of the following:

  * Relapse =< 6 months after first CR, dated from documentation of CR to documentation of relapse
  * Relapse between 6-12 months after first CR
* Refractory to conventional initial induction chemotherapy (=< 2 courses) or to first reinduction (=< 1 course)
* Normal cardiac ejection fraction by pretreatment multi gated acquisition scan (MUGA) or echocardiogram within 4 weeks prior to randomization (resting ejection fraction >= 50% or >= 5% increase with exercise), shortening fraction by echocardiogram >= 24%, or to within the normal range of values for the institution
* Prior treatment to doses of any of the following:

  * < 300 mg/m^2 of doxorubicin
  * < 300 mg/m^2 of daunorubicin
  * < 100 mg/m^2 of idarubicin
  * < 100 mg/m^2 of mitoxantrone
* Serum creatinine =< 2.0 mg/dL
* Serum direct bilirubin < 2.0 mg/dL
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) < 4 x upper limit of normal

  * The above stipulation for normal hepatic function does not apply if liver dysfunction is due to leukemia infiltration
* Prior to study entry, patients must have recovered from toxicities of prior chemotherapy and radiotherapy; for patients refractory to induction chemotherapy (patient subgroup outlined above), marrow documentation of residual leukemia post chemotherapy and qualification for remaining eligibility criteria are needed prior to study entry (this does not require >= 30% marrow blasts to be evident but a minimum of 10% blasts must be present in the marrow)

  * NOTE: Hydroxyurea is permitted within 4 weeks of study entry
* ECOG performance status 0, 1 or 2
* Patients with a history of central nervous system (CNS) leukemia are eligible if there is documentation of no current CNS involvement on cerebrospinal fluid (CSF) examination, (i.e., negative CSF by lumbar puncture)

Consolidation therapy:

* Patients must have an ECOG performance status 0, 1 or 2
* Patients must have documented CR
* Patients must have an absence of infection or have infection controlled by antibiotics; patients who are septic will be excluded
* Patients must have a serum creatinine clearance > 50 cc/minute
* Patients must have a serum direct bilirubin < 2.0 mg/dl and alkaline phosphatase and SGOT (AST) < 4 x upper limits of normal
* Patients must have a normal cardiac ejection fraction by MUGA or echocardiogram prior to consolidation (resting ejection fraction >= 50% or >= 5% increase with exercise), shortening fraction by echocardiogram >= 24%, or to within normal range of values for the institution prior to the first and second cycle of consolidation for arms B and C

Exclusion Criteria

Induction therapy:

* Patients who have relapsed > 1 year after achieving first CR or are in >= second relapse
* Patients who have had a prior allogeneic OR autologous stem cell transplant
* History of recent myocardial infarction (within three months), uncontrolled congestive heart failure, or uncontrolled cardiac arrhythmia
* Prior treatment with carboplatin, topotecan, flavopiridol, or sirolimus
* Pregnant or breast feeding. Women of childbearing potential and sexually active males should use an accepted and effective method of contraception
* Intercurrent organ damage or medical problems that would prohibit therapy; no active or unresolved infection
* Current evidence of invasive fungal infection; such evidence includes positive blood or deep tissue cultures or stains
* Have another (i.e., prior) tumor which is currently active and likely to interfere with the patient's treatment for AML or which is likely to compromise the patient's morbidity or mortality substantially

Consolidation therapy:

* Intercurrent organ damage or medical problems that will jeopardize the outcome of therapy
* For arms B and C, patients have exceeded the following anthracycline doses or their equivalents:
* < 300 mg/m^2 of doxorubicin
* < 300 mg/m^2 of daunorubicin
* < 100 mg/m^2 of idarubicin
* < 100 mg/m^2 of mitoxantrone

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2008-10; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Litzow, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (20):
- United States (19):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - Siouxland Hematology Oncology Associates, Sioux City, Iowa
  - Johns Hopkins University/Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - The Jewish Hospital, Cincinnati, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Geisinger Wyoming Valley, Wilkes-Barre, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
- Rambam Medical Center, Haifa, Israel

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was activated on October 16, 2008 and closed on August 2, 2013 with a total of 92 patients accrued. Duration the response evaluation after meeting the first stage accrual goal, Arm C did not meet the criteria to continue onto the second stage and was closed to accrual at that time.
Groups:
- Arm B (Alvocidib, Mitoxantrone Hydrochloride, Cytarabine): Patients receive alvocidib IV over 4.5 hours qd on days 1-3, cytarabine IV continuously over 72 hours on days 6-8, and mitoxantrone hydrochloride IV over 1-2 hours on day 9.
  alvocidib: Given IV
  mitoxantrone hydrochloride: Given IV
  cytarabine: Given IV
- Arm C (Mitoxantrone Hydrochloride, Cytarabine, Sirolimus): Patients receive sirolimus PO qd on days 2-9, mitoxantrone hydrochloride IV over 15 minutes qd, etoposide IV over 1 hour qd, and cytarabine IV over 3 hours qd on days 4-8 or 5-9. (Closed to accrual)
  mitoxantrone hydrochloride: Given IV
  cytarabine: Given IV
  sirolimus: Given PO
  etoposide: Given IV
Period: Overall Study
Arm/Group | Arm A (Carboplatin and Topotecan Hydrochloride) | Arm B (Alvocidib, Mitoxantrone Hydrochloride, Cytarabine) | Arm C (Mitoxantrone Hydrochloride, Cytarabine, Sirolimus)
Started | 35 | 37 | 20
Eligible and Treated | 35 | 36 | 20
Completed | 34 | 24 | 20
Not Completed | 1 | 13 | 0
Not completed — Never started treatment | 0 | 1 | 0
Not completed — Death | 1 | 6 | 0
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Disease progression/relapse | 0 | 1 | 0
Not completed — Other complicating disease | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Groups:
- Arm A (Carboplatin+Topotecan Hydrochloride): Patients receive carboplatin and topotecan hydrochloride IV continuously over 24 hours on days 1-5.
- Arm B (Alvocidib+Cytarabine+Mitoxantrone): Patients receive alvocidib IV over 4.5 hours qd on days 1-3, cytarabine IV continuously over 72 hours on days 6-8, and mitoxantrone hydrochloride IV over 1-2 hours on day 9.
- Arm C (Sirolimus+Mitoxantrone+Etoposide+Cytarabine): Patients receive sirolimus PO qd on days 2-9, mitoxantrone hydrochloride IV over 15 minutes qd, etoposide IV over 1 hour qd, and cytarabine IV over 3 hours qd on days 4-8 or 5-9. (Closed to accrual)
- Total: Total of all reporting groups
Arm/Group | Arm A (Carboplatin+Topotecan Hydrochloride) | Arm B (Alvocidib+Cytarabine+Mitoxantrone) | Arm C (Sirolimus+Mitoxantrone+Etoposide+Cytarabine) | Total
Number analyzed (Participants) | 35 | 36 | 20 | 91
Age, Continuous [Median (Full Range); unit: years] | 55 [23 to 67] | 62 [19 to 69] | 52 [22 to 68] | 57 [19 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 9 | 37
  Male | 21 | 22 | 11 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 4 | 2 | 7
  White | 33 | 30 | 14 | 77
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 1 | 2
Disease status [Number; unit: participants]
  < 6 months after 1st CR | 9 | 11 | 6 | 26
  6-12 mos after 1st CR | 8 | 8 | 3 | 19
  Refractory | 18 | 17 | 10 | 45
  Unknown/Missing | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: The Rate of Complete Remission (CR+CRi)
Description: CR requires: 1. peripheral blood counts: neutrophil count ≥ 1.0 x 10^9/L, platelet count ≥ 100 x 10^9/L, reduced hemoglobin concentration or hematocrit has no bearing on remission status, and leukemic blasts must not be present in the peripheral blood. 2. bone marrow aspirate and biopsy: maturation of all cell lines must be present, ≤ 5% blasts, auer rods must not be detectable. 3. extramedullary leukemia, such as central nervous system (CNS) or soft tissue involvement, must not be present. CRi requires that all criteria for complete remission be satisfied except patients can have residual neutropenia (<1 x 10^9/L) or thrombocytopenia (<100 x 10^9/L).
Time Frame: Assessed every 3 months for the first 2 years and then every 6 months until relapse or death up to 3 years from registration.
Population: Eligible and treated
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Carboplatin+Topotecan Hydrochloride) | Arm B (Alvocidib+Cytarabine+Mitoxantrone) | Arm C (Sirolimus+Mitoxantrone+Etoposide+Cytarabine)
Number analyzed (Participants) | 35 | 36 | 20
proportion of participants | 0.143 [0.071 to 0.347] | 0.278 [0.161 to 0.43] | 0.15 [0.042 to 0.344]

2. Secondary Outcome: The Rate of Treatment Failure
Description: The definition of treatment failure will include:
  * ≥ 5% leukemic blasts at the time of pre-consolidation marrow
  * Death during/following induction chemotherapy (pre-consolidation)
  * Persisting marrow hypoplasia and pancytopenia for ≥ 2 months after chemotherapy
  * CNS or extramedullary disease at the time of pre-consolidation
  * Leukemia persistence after completion of induction treatment. Leukemia persistence is defined as greater than 10% residual blasts on marrow biopsy done 5-7 days after completion of induction chemotherapy
Time Frame: as for outcome 1
Population: Eligible and treated
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Carboplatin+Topotecan Hydrochloride) | Arm B (Alvocidib+Cytarabine+Mitoxantrone) | Arm C (Sirolimus+Mitoxantrone+Etoposide+Cytarabine)
Number analyzed (Participants) | 35 | 36 | 20
proportion of participants | 0.86 [0.72 to 0.94] | 0.72 [0.57 to 0.84] | 0.84 [0.64 to 0.96]

ADVERSE EVENTS:
Time Frame: Assessed every while on treatment and for 30 days after the end of treatment
Arm/Group | Arm A (Carboplatin+Topotecan Hydrochloride) | Arm B (Alvocidib+Cytarabine+Mitoxantrone) | Arm C (Sirolimus+Mitoxantrone+Etoposide+Cytarabine)
Serious Adverse Events (participants affected / at risk) | 35/35 | 36/36 | 20/20
Other Adverse Events (participants affected / at risk) | 35/35 | 36/36 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Carboplatin+Topotecan Hydrochloride) (N=35) | Arm B (Alvocidib+Cytarabine+Mitoxantrone) (N=36) | Arm C (Sirolimus+Mitoxantrone+Etoposide+Cytarabine) (N=20)
Anemia (Blood and lymphatic system disorders) | 22 | 27 | 11
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 7 | 8 | 11
Hemolysis (Blood and lymphatic system disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1
Death NOS (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 5 | 2
Multi-organ failure (General disorders) | 0 | 3 | 0
Pain (General disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 8 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 4 | 2 | 0
Nausea (Gastrointestinal disorders) | 3 | 4 | 3
Oral hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0
Typhlitis (Gastrointestinal disorders) | 2 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2 | 3
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 1 | 1
Catheter related infection (Infections and infestations) | 4 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 2 | 1 | 1
Lung infection (Infections and infestations) | 1 | 8 | 0
Sepsis (Infections and infestations) | 1 | 7 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0
Upper respiratory infection (Infections and infestations) | 0 | 1 | 0
Infections and infestations - Other (Infections and infestations) | 2 | 9 | 1
Activated PTT prolonged (Investigations) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0
Alkaline phosphatase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 1
Blood bilirubin increased (Investigations) | 2 | 4 | 0
Creatinine increased (Investigations) | 1 | 2 | 0
Fibrinogen decreased (Investigations) | 0 | 1 | 0
GGT increased (Investigations) | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 10 | 16 | 7
Neutrophil count decreased (Investigations) | 34 | 32 | 19
Platelet count decreased (Investigations) | 35 | 36 | 20
Weight loss (Investigations) | 0 | 2 | 0
White blood cell decreased (Investigations) | 35 | 36 | 20
Investigations - Other, specify (Investigations) | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 7 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 7 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 8 | 9 | 1
Hyponatremia (Metabolism and nutrition disorders) | 4 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 9 | 2
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 | 3 | 0
Metabolism and nutrition - Other (Metabolism and nutrition disorders) | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Dysphasia (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Nervous system disorders - Other (Nervous system disorders) | 0 | 1 | 0
Blurred vision (Eye disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Renal and urinary disorders - Other (Renal and urinary disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 5 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Carboplatin+Topotecan Hydrochloride) (N=35) | Arm B (Alvocidib+Cytarabine+Mitoxantrone) (N=36) | Arm C (Sirolimus+Mitoxantrone+Etoposide+Cytarabine) (N=20)
Anemia (Blood and lymphatic system disorders) | 34 | 32 | 20
Sinus tachycardia (Cardiac disorders) | 0 | 4 | 2
Chills (General disorders) | 1 | 10 | 4
Edema limbs (General disorders) | 5 | 8 | 4
Fatigue (General disorders) | 16 | 12 | 9
Fever (General disorders) | 5 | 2 | 0
Pain (General disorders) | 0 | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 6 | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 9 | 4
Abdominal pain (Gastrointestinal disorders) | 3 | 3 | 1
Constipation (Gastrointestinal disorders) | 3 | 6 | 2
Diarrhea (Gastrointestinal disorders) | 21 | 23 | 13
Dry mouth (Gastrointestinal disorders) | 1 | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 2 | 1
Mucositis oral (Gastrointestinal disorders) | 7 | 11 | 7
Nausea (Gastrointestinal disorders) | 18 | 18 | 9
Oral pain (Gastrointestinal disorders) | 2 | 1 | 0
Vomiting (Gastrointestinal disorders) | 10 | 10 | 4
Cytokine release syndrome (Immune system disorders) | 0 | 2 | 0
Infections and infestations - Other (Infections and infestations) | 0 | 3 | 0
Alanine aminotransferase increased (Investigations) | 14 | 12 | 4
Alkaline phosphatase increased (Investigations) | 12 | 14 | 8
Aspartate aminotransferase increased (Investigations) | 15 | 16 | 5
Blood bilirubin increased (Investigations) | 2 | 14 | 4
Creatinine increased (Investigations) | 4 | 9 | 2
ECG QT corrected interval prolonged (Investigations) | 1 | 2 | 0
INR increased (Investigations) | 0 | 2 | 1
Lymphocyte count decreased (Investigations) | 3 | 0 | 0
Neutrophil count decreased (Investigations) | 18 | 13 | 12
Platelet count decreased (Investigations) | 26 | 24 | 17
Weight loss (Investigations) | 3 | 3 | 2
White blood cell decreased (Investigations) | 24 | 18 | 16
Investigations - Other, specify (Investigations) | 1 | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 12 | 8 | 6
Hyperglycemia (Metabolism and nutrition disorders) | 10 | 14 | 8
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypernatremia (Metabolism and nutrition disorders) | 2 | 3 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 3 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 9 | 11 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 9 | 10 | 5
Hypokalemia (Metabolism and nutrition disorders) | 4 | 9 | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 7 | 4
Hyponatremia (Metabolism and nutrition disorders) | 6 | 6 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 4 | 5 | 4
Metabolism and nutrition - Other (Metabolism and nutrition disorders) | 4 | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Dizziness (Nervous system disorders) | 0 | 3 | 1
Dysgeusia (Nervous system disorders) | 3 | 4 | 3
Headache (Nervous system disorders) | 5 | 5 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 1 | 0
Insomnia (Psychiatric disorders) | 3 | 4 | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 6 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Urinary frequency (Renal and urinary disorders) | 1 | 2 | 0
Hematoma (Vascular disorders) | 1 | 2 | 0
Hypertension (Vascular disorders) | 2 | 0 | 0
Hypotension (Vascular disorders) | 9 | 6 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less